CLINICAL TRIAL: NCT06184178
Title: Implementing the Transcultural Social-Ethical-Care Model -TEC-MED for Older People in the Mediterranean Basin
Acronym: TEC-MED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: REGINA ALLANDE CUSSO (Other)
Responsible Party: Sponsor-Investigator, REGINA ALLANDE CUSSO, Clinical Professor, University of Seville
Organization: University of Seville (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: A_A 3 2_0376; TEC-MED (Other: University of Seville)
Record Dates: First submitted 2023-12-05; First posted 2023-12-28 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Older People; Care Dependency; Social Exclusion
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTERVENTION GROUP (Experimental): Implementation of socio-health care based on TEC-MED model
  Interventions: Other: Socio-health care
- CONTROL GROUP (No Intervention): No intervention

INTERVENTIONS:
Other: Socio-health care — Socio-health care under TEC-MED model and an integral assessment
  Other Names: TEC-MED care model
  Arms: INTERVENTION GROUP

SUMMARY:
Implementation of the TEC-MED model of social and health care in the elderly population of the Mediterranean basin through a quasi-experimental trial. Participants will be assigned to the intervention group and will receive comprehensive care and assessment under the TEC-MED care model. Participants in the control group will receive usual care during the data collection phase, but will be offered care under the TEC-MED model at the end of the project.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or more
* Living in the Mediterranean Basin countries

Exclusion Criteria:

* None

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20000 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Care Dependency Level | 3 months
  Assessment of the care dependency level using INICIARE Scale. The scale measures the care dependency level, framed in three levels: low level, mid level, high level. The expected outcome is to mantain the care dependency level, or low level, from the fisrt assessment to the second.

SECONDARY OUTCOMES:
Quality of life level | 3 months
  Assessment of the quality of life level, using the EQ-5D-5L Scale. The scale measures the quality of life level, framed in two levels: low level and high level. The expected outcome is to improve the quality of live level, from the fisrt assessment to the second.

CONTACTS AND LOCATIONS:
Overall Officials: Regina Allande-Cussó, Dr., Study Director — University of Seville
Locations (1):
- University of Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: No
All personal data will be kept under confidentiality

REFERENCES:
- [Derived] Lima-Serrano M, Allande-Cusso R, Vargas-Martinez AM, Karam G, El-Korh L, Porcel-Galvez AM. Testing the TEC-MED-Integrated Transcultural Social-Ethical-Care Model for Older People in the Mediterranean Basin: A Mixed-Method Quasiexperimental Study Protocol. Int J Integr Care. 2025 May 9;25(2):9. doi: 10.5334/ijic.9017. eCollection 2025 Apr-Jun. PMID 40352956
- See also: Webpage of the project — https://www.enicbcmed.eu/projects/tec-med